CLINICAL TRIAL: NCT05442021
Title: Impact of Direct Current Neuromuscular Electrical Stimulation on Physical Therapy Treatment of Peripheral Neuropathy
Brief Title: Direct Current Neuromuscular Electrical Stimulation for Treatment of Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuFit - Neurological Fitness and Education (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00063515
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Neuropathy
Keywords: electrical stimulation; neubie; neuromuscular electrical stimulation
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Study will be divided into two randomly assigned groups - control and experimental. Control group will receive traditional e-stim treatment with TENS plus physical therapy. Experimental group will receive direct current e-stim treatment with the Neubie device plus physical therapy.
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be assessed by clinicians at Hands on Diagnostics locations. Assessors will be blinded to which intervention participant has received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Neubie Direct Current Electrical Stimulation (Experimental): The experimental group subjects follow with 12 sessions of physical therapy over a 6-week period which include: a 30-min foot bath session using the Neubie and 15-min of various physical therapy exercises.
  Interventions: Device: Neubie Direct Current Electrical Stimulation Device
- Transcutaneous Electrical Nerve Stimulation (Other): The control group subjects follow with 12 sessions of physical therapy over a 6-week period which include: a 30-min footbath with TENS and 15-min of various physical therapy exercises.
  Interventions: Device: TENS

INTERVENTIONS:
Device: Neubie Direct Current Electrical Stimulation Device — Direct Current Electrical Stimulation Device that uses electrodes non-invasively on the skin to stimulate muscle fibers.
  Arms: Neubie Direct Current Electrical Stimulation
Device: TENS — Transcutaneous Electrical Nerve Stimulation device - uses alternating current delivered through electrodes on the skin.
  Arms: Transcutaneous Electrical Nerve Stimulation

SUMMARY:
This study will compare two methods of electrical stimulation (alternating current and direct current) as an adjunctive therapy to treating peripheral neuropathy. Both types of electrical stimulation have been used in clinical practice for physical therapy, however direct current stimulation is much less common and there is less known about their impact on physical therapy outcomes. The aim of this project is to show the efficacy of a novel device, the Neubie direct current device, compared to traditional TENS unit, in clinical physical therapy treatment of neuropathy. Outcomes measured will include three methods of two-point discrimination, vibration sense, pain, and score on the modified Toronto Clinical Neuropathy scale.

DETAILED DESCRIPTION:
To determine the efficacy of direct current electrical stimulation (the Neubie device) on long-term symptoms and severity of neuropathy, participants will enroll in a 6-week treatment regimen at one of 9 Hands On Physical Therapy associated clinic sites listed included in application. The first session will consist of an EMG/NCS evaluation to determine severity of neuropathy and to rule out polyneuropathy, which will serve as baseline (and a within subject control) for the intervention.

Participants will then undergo a specialized neuropathy protocol that includes traditional PT therapy for neuropathy, as well as treatment with the Neubie (or traditional e-stim) both during PT exercises and as additional treatment after sessions. Subjects receive an evaluation session that includes an Electrodiagnostic Study, pain assessment, evaluation of two-point discrimination, and vibration sense.

The experimental group subjects follow with 12 sessions of physical therapy over a 6-week period which include: a 30-min foot bath session with the Neubie and 15-min of various physical therapy exercises.

The control group subjects follow with 12 sessions of physical therapy over a 6-week period which include: a 30-min footbath with TENS and 15-min of various physical therapy exercises.

At the end of the 12 sessions of treatment, subjects receive a final evaluation session that includes an Electrodiagnostic Study, pain assessment, evaluation of two-point discrimination, and vibration sense.

Participants will receive 12 treatments over 6 weeks. EMG/NCS and a neuropathy pain questionnaire will be measured at both the initial evaluation and at the completion of the final session, and will provide both quantitative and qualitative data on the severity of neuropathy symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Must have a minimum score of 1 on the modified Toronto Clinical Neuropathy Score
* Must be able to attend weekly sessions for the 6 week period of the study (no extended travel)
* Must be at least 18 years old.

Exclusion Criteria:

* Currently pregnant
* Cardiac pacemaker
* Active or recent cancer in the lower limbs
* Active or recent blood clots in the lower limbs
* History of epilepsy
* No open wounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Distal Latency | Pre-intervention
  The time in milliseconds that it takes the impulse to travel from the stimulation point at the wrist to the recording electrode.
Distal Latency | 6 weeks
  The time in milliseconds that it takes the impulse to travel from the stimulation point at the wrist to the recording electrode.
Tibial Motor Nerve Conduction Velocity | Pre-intervention
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the Tibial Motor Nerve.
Tibial Motor Nerve Conduction Velocity | 6 weeks
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the Tibial Motor Nerve.
Fibular Motor Nerve Conduction Velocity | 6 weeks
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the Fibular Motor Nerve.
Fibular Motor Nerve Conduction Velocity | Pre-intervention
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the Fibular Motor Nerve.
Ulnar Motor Nerve Conduction Velocity | Pre-intervention
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the Ulnar Motor Nerve.
Ulnar Motor Nerve Conduction Velocity | 6 weeks
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the Ulnar Motor Nerve.
Sural Sensory Nerve Conduction Velocity | Pre-intervention
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the Sural Sensory Nerve.
Sural Sensory Nerve Conduction Velocity | 6 weeks
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the Sural Sensory Nerve.
Superficial Fibular Sensory Nerve Conduction Velocity | 6 weeks
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the Superficial Fibular Sensory Nerve.
Superficial Fibular Sensory Nerve Conduction Velocity | Pre-intervention
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the Superficial Fibular Sensory Nerve.
Ulnar Sensory Nerve Conduction Velocity | Pre-intervention
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the Ulnar Sensory Nerve.
Ulnar Sensory Nerve Conduction Velocity | 6 weeks
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the Ulnar Sensory Nerve.
Tibial F-Wave | Pre-intervention
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the Tibial F-Wave.
Tibial F-Wave | 6 weeks
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the Tibial F-Wave.
H-Reflex | 6 weeks
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the H-Reflex.
H-Reflex | Pre-intervention
  Electrodes on the skin release tiny electric shocks to stimulate nerves; the amplitude of the nerve signal will be measured for the H-Reflex.

CONTACTS AND LOCATIONS:
Overall Officials: Ramona von Leden, PhD, Study Director — NeuFit - Neurological Fitness and Education
Locations (11):
- United States (11):
  - APEX Physical Therapy, Cape Coral, Florida
  - Catalyst Physical Therapy, Clearwater, Florida
  - APEX Physical Therapy, Fort Myers, Florida
  - Diagnostic Solutions, Springfield, Kentucky
  - Hands-On Physical Therapy, Astoria, New York
  - Hands-On Physical Therapy of Queens Village, Queens Village, New York
  - Panetta Physical Therapy & Diagnostics, Ronkonkoma, New York
  - Courcier Physical Therapy, Edmond, Oklahoma
  - Spine & Rehab Specialists, El Paso, Texas
  - Active Fitness Physical Therapy, Oak Hill, West Virginia
  - Active Fitness Physical Therapy, Victor, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Snyder MJ, Gibbs LM, Lindsay TJ. Treating Painful Diabetic Peripheral Neuropathy: An Update. Am Fam Physician. 2016 Aug 1;94(3):227-34. PMID 27479625
- [Background] Rogers LC, Andros G, Armstrong DG. Update from the Diabetic Foot Global Conference (DFCon) 2007. Int Wound J. 2007 Dec;4(4):295-7. doi: 10.1111/j.1742-481X.2007.00377.x. No abstract available. PMID 18154623
- [Background] Thakral G, Kim PJ, LaFontaine J, Menzies R, Najafi B, Lavery LA. Electrical stimulation as an adjunctive treatment of painful and sensory diabetic neuropathy. J Diabetes Sci Technol. 2013 Sep 1;7(5):1202-9. doi: 10.1177/193229681300700510. PMID 24124947
- [Background] Ziegler D. Treatment of diabetic polyneuropathy: Update 2006. Ann N Y Acad Sci. 2006 Nov;1084:250-66. doi: 10.1196/annals.1372.008. PMID 17151306
- [Background] Sluka KA, Walsh D. Transcutaneous electrical nerve stimulation: basic science mechanisms and clinical effectiveness. J Pain. 2003 Apr;4(3):109-21. doi: 10.1054/jpai.2003.434. PMID 14622708
- [Background] Peters EJ, Armstrong DG, Wunderlich RP, Bosma J, Stacpoole-Shea S, Lavery LA. The benefit of electrical stimulation to enhance perfusion in persons with diabetes mellitus. J Foot Ankle Surg. 1998 Sep-Oct;37(5):396-400; discussion 447-8. doi: 10.1016/s1067-2516(98)80048-3. PMID 9798171
- [Background] Gilcreast DM, Stotts NA, Froelicher ES, Baker LL, Moss KM. Effect of electrical stimulation on foot skin perfusion in persons with or at risk for diabetic foot ulcers. Wound Repair Regen. 1998 Sep-Oct;6(5):434-41. doi: 10.1046/j.1524-475x.1998.60505.x. PMID 9844163
- [Background] da Silva MP, Liebano RE, Rodrigues VA, Abla LE, Ferreira LM. Transcutaneous electrical nerve stimulation for pain relief after liposuction: a randomized controlled trial. Aesthetic Plast Surg. 2015 Apr;39(2):262-9. doi: 10.1007/s00266-015-0451-6. Epub 2015 Feb 10. PMID 25665520
- [Background] Ordog GJ. Transcutaneous electrical nerve stimulation versus oral analgesic: a randomized double-blind controlled study in acute traumatic pain. Am J Emerg Med. 1987 Jan;5(1):6-10. doi: 10.1016/0735-6757(87)90281-6. PMID 3545246
- [Background] Zhao M, Bai H, Wang E, Forrester JV, McCaig CD. Electrical stimulation directly induces pre-angiogenic responses in vascular endothelial cells by signaling through VEGF receptors. J Cell Sci. 2004 Jan 26;117(Pt 3):397-405. doi: 10.1242/jcs.00868. Epub 2003 Dec 16. PMID 14679307
- [Background] Kanno S, Oda N, Abe M, Saito S, Hori K, Handa Y, Tabayashi K, Sato Y. Establishment of a simple and practical procedure applicable to therapeutic angiogenesis. Circulation. 1999 May 25;99(20):2682-7. doi: 10.1161/01.cir.99.20.2682. PMID 10338463
- [Background] Reichstein L, Labrenz S, Ziegler D, Martin S. Effective treatment of symptomatic diabetic polyneuropathy by high-frequency external muscle stimulation. Diabetologia. 2005 May;48(5):824-8. doi: 10.1007/s00125-005-1728-0. Epub 2005 Apr 14. PMID 15830180
- [Background] DeSantana JM, Walsh DM, Vance C, Rakel BA, Sluka KA. Effectiveness of transcutaneous electrical nerve stimulation for treatment of hyperalgesia and pain. Curr Rheumatol Rep. 2008 Dec;10(6):492-9. doi: 10.1007/s11926-008-0080-z. PMID 19007541
- [Background] Doucet BM, Griffin L. High-versus low-frequency stimulation effects on fine motor control in chronic hemiplegia: a pilot study. Top Stroke Rehabil. 2013 Jul-Aug;20(4):299-307. doi: 10.1310/tsr2004-299. PMID 23893829
- [Background] Najafi B, Talal TK, Grewal GS, Menzies R, Armstrong DG, Lavery LA. Using Plantar Electrical Stimulation to Improve Postural Balance and Plantar Sensation Among Patients With Diabetic Peripheral Neuropathy: A Randomized Double Blinded Study. J Diabetes Sci Technol. 2017 Jul;11(4):693-701. doi: 10.1177/1932296817695338. Epub 2017 Feb 1. PMID 28627217
- [Background] Chandrasekaran S, Davis J, Bersch I, Goldberg G, Gorgey AS. Electrical stimulation and denervated muscles after spinal cord injury. Neural Regen Res. 2020 Aug;15(8):1397-1407. doi: 10.4103/1673-5374.274326. PMID 31997798
- [Background] Zehr EP, Collins DF, Chua R. Human interlimb reflexes evoked by electrical stimulation of cutaneous nerves innervating the hand and foot. Exp Brain Res. 2001 Oct;140(4):495-504. doi: 10.1007/s002210100857. PMID 11685403
- [Result] Yang, Z. et al. Scoring systems to screen for diabetic peripheral neuropathy. (Cochrane Database Syst Rev. 2018 Jul 30;2018(7):CD010974. doi: 10.1002/14651858.CD010974.pub2. eCollection 2018 Jul.).
- [Derived] Kostopoulos D, Rizopoulos K, McGilvrey J, Hauskey J, Courcier J, Connor-Israel K, Koster H, von Leden R. An Open-Label Comparative Study of the Impact of Two Types of Electrical Stimulation (Direct Current Neuromuscular Electrical Stimulation and Transcutaneous Electrical Stimulation) on Physical Therapy Treatment of Diabetic Peripheral Neuropathy. J Diabetes Res. 2025 Feb 4;2025:9970124. doi: 10.1155/jdr/9970124. eCollection 2025. PMID 39949402